CLINICAL TRIAL: NCT02580773
Title: A Prospective, Randomized, Double-blind, Placebo Controlled, Multi-national Study of Therapeutic Anticoagulation Strategy for Acute Chest Syndrome in Adults
Brief Title: Therapeutic Anticoagulation Strategy for Acute Chest Syndrome
Acronym: TASC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOR14068
Record Dates: First submitted 2015-10-05; First posted 2015-10-20 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2020-04

CONDITIONS: Anemia; Sickle Cell; Acute Chest Syndrome; Low-Molecular-Weight Heparin
Keywords: Sickle cell disease; Anemia; Rare disease; Reanimation; Prophylactic anticoagulation
MeSH Terms: conditions — Anemia; Acute Chest Syndrome; Anemia, Sickle Cell; Rare Diseases | interventions — Tinzaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic anticoagulation (Other)
  Interventions: Drug: Prophylactic anticoagulation ( INNOHEP®)
- Curative anticoagulation (Experimental)
  Interventions: Drug: Curative anticoagulation ( INNOHEP®)

INTERVENTIONS:
Drug: Prophylactic anticoagulation ( INNOHEP®) — subcutaneous anticoagulation with low molecular weight heparin (tinzaparin) at a prophylactic dose (4500 UI/day)
  Arms: Prophylactic anticoagulation
Drug: Curative anticoagulation ( INNOHEP®) — subcutaneous anticoagulation with low molecular weight heparin (tinzaparin) at a curative dose (175 UI/kg/day for 7 days)
  Arms: Curative anticoagulation

SUMMARY:
Acute Chest Syndrome (ACS) is a pulmonary complication of sickle cell disease (SCD) representing the leading cause of death and the second cause of hospitalization among adult patients. Pulmonary vaso-occlusion is one of the main pathophysiologic hypotheses during ACS. Our hypothesis is that therapeutic anticoagulation may reduce the severity of ACS via the alleviation of pulmonary thrombosis. The main objective of this prospective, randomized, double-blind study is to test the efficacy and safety of a curative anticoagulation strategy during ACS. The main efficacy endpoint is time to ACS resolution. The main safety endpoint is number of major bleedings.

A thoracic CT scan will be performed to check for pulmonary artery thrombosis. If the CT scan is positive (thrombosis within a large elastic artery), the patient will not be randomized and will be treated with a curative anticoagulation. If the CT scan is negative, the patient will be randomized to receive subcutaneous anticoagulation with low molecular weight heparin (tinzaparin) either at a curative dose (175 Unit International (UI)/kg/day for 7 days) or at a prophylactic dose (4500 UI/day).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Major sickle cell syndrome (SS, SC, Sβ)
* ACS defined by the association of a new infiltrate on chest X-ray or CT scan and a respiratory symptom or abnormal chest auscultation
* Written, informed consent

Main Exclusion Criteria:

* Pregnancy, post-partum
* Iodine allergy
* Extreme weight (<40 kg or > 100 kg)
* Moderate to severe renal insufficiency
* Moya-moya disease
* Symptomatic cerebral aneurysm
* Major transfusional risk
* Uncontrolled severe retinopathy
* All other contra-indications to curative anti-coagulation by tinzaparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
The main efficacy endpoint is time to ACS resolution | up to 15 days
  The delay between randomization and ACS resolution
Number of major bleedings | up to 15 days

SECONDARY OUTCOMES:
Number of complicated ACS | up to 15 days
Blood volume exchanged | up to 15 days
Cumulative dose of opioids | up to 15 days
Hospital mortality | up to 15 days
Duration of hospital stay | up to 15 days
Number of non-major bleedings | up to 15 days
Number of readmissions and thromboembolic events within 6 months | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Maitre, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Armand Mekontso Dessap, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Qari MH, Aljaouni SK, Alardawi MS, Fatani H, Alsayes FM, Zografos P, Alsaigh M, Alalfi A, Alamin M, Gadi A, Mousa SA. Reduction of painful vaso-occlusive crisis of sickle cell anaemia by tinzaparin in a double-blind randomized trial. Thromb Haemost. 2007 Aug;98(2):392-6. PMID 17721622
- [Background] Mekontso Dessap A, Deux JF, Abidi N, Lavenu-Bombled C, Melica G, Renaud B, Godeau B, Adnot S, Brochard L, Brun-Buisson C, Galacteros F, Rahmouni A, Habibi A, Maitre B. Pulmonary artery thrombosis during acute chest syndrome in sickle cell disease. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1022-9. doi: 10.1164/rccm.201105-0783OC. PMID 21836136
- [Derived] Mekontso Dessap A, Habibi A, Arlet JB, Fartoukh M, Guerin L, Guillaud C, Roux D, Oziel J, Ngo S, Carpentier B, Lopez-Sublet M, Affo L, Melica G, Etienne-Julan M, Delacroix I, Lionnet F, Loko G, Da Silva D, Michel M, Razazi K, Charles-Nelson A, Bartolucci P, Gendreau S, Katsahian S, Maitre B. Comparison of Prophylactic and Therapeutic Doses of Anticoagulation for Acute Chest Syndrome in Sickle Cell Disease: The TASC Double-Blind Controlled Randomized Clinical Trial. Am J Respir Crit Care Med. 2025 May;211(5):832-841. doi: 10.1164/rccm.202409-1727OC. PMID 40209087